CLINICAL TRIAL: NCT02838836
Title: Tumor Cell and DNA Detection in the Blood, Urine and Bone Marrow of Patients With Solid Cancers
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jussuf Kaifi, Assistant Professor, Chief, Section for Thoracic Surgery, University of Missouri-Columbia
Other Study IDs: 2010166
Record Dates: First submitted 2016-07-09; First posted 2016-07-20 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer; Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Hepatocellular Cancer; Colorectal Cancer
Keywords: Cancer; Circulating tumor cells (CTCs); Disseminated tumor cells (DTCs); Circulating tumor DNA (ctDNA)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Colorectal Neoplasms; Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, bone marrow, tissue, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study sample collection: Blood draws, urine and tissue asservation, and bone marrow aspiration will be done during surgery
  Interventions: Procedure: Study sample collection

INTERVENTIONS:
Procedure: Study sample collection — Blood draws, urine and tissue asservation, and bone marrow aspiration will be done during surgery

SUMMARY:
Patients with resectable solid primary cancers and even limited number of metastases are potentially curable. However, most patients develop recurrences despite surgery. Circulating and disseminated tumor cell (CTC/DTC) and circulating cell-free (cf) DNA isolation from the blood, urine and bone marrow will increase understanding of cancer spread and advance knowledge to develop individualized therapies.

DETAILED DESCRIPTION:
Background:

Patients with resectable solid primary cancers and even limited number of metastases are potentially curable. However, most patients develop recurrences despite surgery. Circulating and disseminated tumor cell (CTC/DTC) and circulating cell-free (cf) DNA isolation from the blood, urine and bone marrow will increase understanding of cancer spread and advance knowledge to develop individualized therapies.

Hypothesis and Rationale:

CTCs/DTCs and cfDNA isolated from the blood, urine and bone marrow during cancer surgeries undergo pheno- and/or genotype changes. CTCs/DTCs have potential for dissemination and tumor growth in vivo. Investigating the biology of liquid biomarkers in the blood, urine and bone marrow will significantly increase understanding of cancer biology.

Specific Aims:

CTCs/DTCs and cfDNA isolated from cancer patients will be characterized for genetic alterations and expression of key signaling/proliferation biomarkers and grow in vivo in nude mice.

Study Design:

100 patients undergoing solid cancer surgeries will be recruited for perioperative CTC/DTC/cfDNA isolation from the blood, urine and bone marrow with innovative techniques. In addition, 20 patients undergoing similar surgeries for benign disease will also be included as controls. CTCs/DTCs, cfDNA and cancer tissue pheno- and/or genotype analysis will be performed with different innovative techniques. Furthermore, CTCs/DTCs will be enriched, cultured and characterized. Tumor growth potential will be studied in nude mice.

Relevance:

This translational cancer trial addresses fundamental aspects of cancer disease being the cause of death in 1 out of 4 persons in the US. Innovative CTCs/DTCs characterization can shed light on the tumor biology, and identify therapy targets. Results of this study can be fundamentally important to understanding cancer spread and development of personalized therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years.
* Subjects of all genders and ethnicities.
* Subjects with the diagnosis of a solid cancer (n=100) of all stages will be included (lung, esophageal, stomach, bile duct/pancreas, colorectal, melanoma, sarcoma).
* Ten patients with no present suspicion and no previous history of any cancer (except basal cell cancer of the skin) that undergo surgeries for other benign indications will serve as controls (n=20).
* In patients undergoing surgery for cancer the histopathology should preferably be pathologically proven by a previous or novel biopsy. Yet, patients with a high cancer suspicion by radiology and clinical picture that undergo cancer surgery will not be excluded. No additional biopsies, testing or interventions will be performed for the purpose of this study if the medical treatment will not require it.
* Subjects must be capable of giving informed consent.

Exclusion Criteria:

* Pregnant women.
* Subjects with the concurrent diagnosis of an active secondary (synchronous) malignancy besides basal cell carcinoma of the skin will be excluded, if there is evidence of disease burden or if the patient is currently being treated with chemotherapy.
* Subjects with a hemoglobin of <8g/dl in the morning of the procedure will be excluded.
* In subjects who require intraoperative transfusions of >4 units of red packed blood cells (RPBCs), no further blood will be drawn for CTC/DTC/cfDNA analysis during surgery or on postoperative day 1.
* In patients with coagulation disorders that could lead to significant bleeding (such as hemophilia, significant thrombocytopenia) requiring prophylactic administration of coagulative products, no bone marrow aspiration will be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with the diagnosis of a solid cancer of all stages will be included (lung, esophageal, stomach, bile duct/pancreas, colorectal, melanoma, sarcoma).
Sampling Method: Non-Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
CTC/DTC numbers measured in blood, urine and bone marrow samples will be correlated with patient outcome | 5 years
  CTC/DTC numbers in the blood, urine and bone marrow will be determined and correlated with survival data (presence of recurrence, death) by univariate analysis (log rank test), multivariate analysis (Cox regression) and t test/ANOVA

SECONDARY OUTCOMES:
ctDNA characteristics will be correlated with survival data | 5 years
  A panel of ctDNA mutations detected in the blood will be gathered in a score and correlated with survival data (presence of recurrence, death) by univariate analysis (log rank test), multivariate analysis (Cox regression)

CONTACTS AND LOCATIONS:
Overall Officials: Jussuf T Kaifi, MD, PhD, Principal Investigator — Ellis Fischel Cancer Center, University of Missouri
Locations (1):
- Ellis Fischel Cancer Center, University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suvilesh KN, Nussbaum YI, Radhakrishnan V, Manjunath Y, Avella DM, Staveley-O'Carroll KF, Kimchi ET, Chaudhuri AA, Shyu CR, Li G, Pantel K, Warren WC, Mitchem JB, Kaifi JT. Tumorigenic circulating tumor cells from xenograft mouse models of non-metastatic NSCLC patients reveal distinct single cell heterogeneity and drug responses. Mol Cancer. 2022 Mar 12;21(1):73. doi: 10.1186/s12943-022-01553-5. PMID 35279152

DOCUMENTS (1):
  • Informed Consent Form (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT02838836/ICF_000.pdf